CLINICAL TRIAL: NCT07146516
Title: Ora Secunda Cerclage Laser Retinopexy To Prevent Retinal Detachment In Stickler Syndrome (OSC/SS): A Prospective Historically Controlled Study
Brief Title: Retinal Detachment Prevention (Laser Prophylaxis) in Stickler Syndrome (SS)
Acronym: OSC/SS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller Eye Research Foundation (Other)
Collaborators: Five Lakes Clinical Research Consulting, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSC/SS
Record Dates: First submitted 2025-07-03; First posted 2025-08-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Stickler Syndrome Type 1; Stickler Syndrome Type 2
Keywords: prophylactic laser retinopexy; Ora Secunda Cerclage; laser; prophylactic; retinopexy; Stickler syndrome; retinal detachment; retinal tear; Stickler syndrome type 2; giant retinal tear; encircling laser prevention; Stickler syndrome type 1; GRT
MeSH Terms: conditions — Stickler syndrome, type 1; Stickler syndrome, type 2; Retinal Detachment; Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children, Adolescents, and Adults with SS treated with Prophylactic Laser Retinopexy (Experimental): Intervention: Children, Adolescents, and Adults with SS treated with prophylactic laser retinopexy procedure.
  Interventions: Procedure: Prophylactic (non-invasive) Laser Retinopexy

INTERVENTIONS:
Procedure: Prophylactic (non-invasive) Laser Retinopexy — Prophylactic laser retinopexy to prevent RD in participants with SS using the indirect ophthalmoscopy (IDO) to place approximately 1500 to 2500 moderate intensity burns to produce encircling grid pattern, placed one burn width apart from 2 MM anterior to the ora serrata, extending to and between the vortex vein ampullae.

SUMMARY:
The goal of this clinical trial is to prospectively document to what extent the OSC/SS prophylactic laser retinopexy procedure works to prevent retinal detachment in SS in children and adults.

Researchers will compare the OSC/SS procedure in SS to the natural progression of SS to see to what extent the OSC/SS procedure works to prevent retinal detachment.

Participants will:

* Have the OSC/SS procedure in one or both eyes
* Have eye tests
* Have genetic testing for SS as needed
* Visit the study center 9 times over 5 years for checkups and tests

DETAILED DESCRIPTION:
Prophylactic treatment for RD has been well-documented to be safe and effective for specific predisposing conditions, but parameters are not standardized and are poorly documented in the literature for Stickler syndrome. There is significant, but only retrospective, evidence in the scientific literature that non-invasive, encircling (360 degree) laser prophylaxis (cerclage prophylaxis) reduces the rate of retinal detachment in patients with Stickler syndrome by approximately five-fold. In February 2025, the American Academy of Ophthalmology (AAO) endorsed 360-degree cerclage laser prophylaxis for Stickler syndrome based on retrospective evidence. A statistical review of pertinent articles concluded that prophylactic laser therapy was associated with a significantly lower risk of retinal detachment in patients with Stickler syndrome compared to no laser prophylaxis. This clinical trial is designed to offer OSC/SS as the optimal form of such prevention, and to prospectively document, in a standardized manner, the extent to which it prevents retinal detachment in patients with Stickler syndrome.

This clinical trial aims to address the lack of standardized documentation in previous literature and studies by providing standardized treatment parameters and rigorously documenting the OSC/SS technique. By evaluating the safety and efficacy of OSC/SS in preventing RD in Stickler syndrome patients, this study seeks to establish a benchmark for future clinical practice and research.

The primary objective is to demonstrate the efficacy of the OSC/SS procedure compared to the natural progression of SS to prevent RD for individuals with SS. This comparison will be made using historical control data provided by Cambridge University, which documents the rate of occurrence of RD in the absence of prior prophylactic treatment. Cambridge University maintains a large SS database, consisting of decades of clinical and research data on Stickler syndrome populations, providing the necessary control raw data for this study population. If the OSC/SS procedure proves to be adequately successful in the study, then it may become the gold standard treatment used to prevent RD in patients with SS and, with modifications, other populations at high risk for RD.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for prophylactic laser retinopexy
2. Capable of giving signed informed consent, and assent (as appropriate)
3. Signature of research informed consent form from participant, or participant's legally authorized representative (LAR)/parent(s)/legal guardian
4. Male or female of any age
5. SS type 1 or type 2 confirmed by genetic testing

Exclusion Criteria:

1. Presence of media opacity (for example, dense cataract, corneal scar) or poor pupillary dilation that precludes adequate OSC/SS performance, laser treatment, or imaging.
2. Prior prophylactic laser treatment that cannot be supplemented to achieve a complete OSC/SS pattern or exceeds the designated OSC/SS pattern.
3. RD in the eye to be treated.
4. Significant intraocular hemorrhage in the eye to be treated.
5. Uncontrolled ocular conditions (e.g., glaucoma) that may be worsened by the procedure or preclude follow-up.
6. Any other ocular condition that precludes the ability to perform adequate laser treatment under scleral depression.
7. Any systemic medical contraindication where the risk of intervention outweighs the potential benefit.
8. Known pathogenic mutations in genes associated with other inherited retinal detachment syndromes, including but not limited to: FEVR-related genes: FZD4, LRP5, TSPAN12, NDPX-linked retinoschisis (RS1) Wagner Syndrome (VCAN).
9. Other syndromes associated with increased risk of retinal detachment (for example, Knobloch syndrome, Marfan syndrome, Pierson syndrome).
10. History of Coats disease.
11. History of Retinopathy of Prematurity (with or without laser treatment).
12. Previous laser photocoagulation in the study eye for any indication, including Retinopathy of prematurity (ROP) Panretinal photocoagulation for diabetic retinopathy.
13. Laser to lattice degeneration or 360-degree laser cerclage for Stickler Syndrome that cannot be supplemented to meet OSC/SS criteria.
14. Previous cryopexy.
15. Previous scleral buckle.
16. Previous vitrectomy in the study eye for any reason.
17. Significant peripheral retinal pathology unrelated to Stickler that increases the risk of retinal detachment including but not limited to: retinoschisis, hemorrhages, angiomatous lesions, pars planitis.
18. History of ocular trauma with significant trauma to the posterior segment of the eye and may increase the risk of retinal detachment including Ruptured globe, Vitreous hemorrhage, Commotio retinae, Traumatic macular hole, Intraocular foreign body.
19. Inability or unwillingness to comply with required follow-up schedule (clinical visits, imaging).
20. Anticipated relocation, foster care instability, or any factor significantly limiting longitudinal follow-up.
21. Investigator judgment: Any condition not listed above that could interfere with the trial's integrity or subject safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with SS who Develop RD After Undergoing the OSC/SS Procedure as Assessed by One of the Following Photographic Fundus Mapping and IDO Examinations | From enrollment to post initial procedure at 5 years
  Efficacy of the OSC/SS procedure in preventing RD in participants with type 1 (STL1) and type 2 (STL2) SS will be assessed annually by tracking the number of participants who develop RD after undergoing the OSC/SS procedure, using data from one of the following: photographic fundus mapping and IDO examinations.

SECONDARY OUTCOMES:
Frequency of Adverse Events as Assessed by Recurring Eye Evaluations (photographic fundus mapping, OCT, intraocular pressure, pupil measurements, slit lamp biomicroscopy, motility assessments, and vision acuity testing) | From enrollment to post initial procedure at 5 years
  Annual evaluation of the safety of the OSC/SS procedure will be assessed by reviewing adverse events collected from recurring visual history and eye evaluations (photographic fundus mapping, OCT, intraocular pressure, pupil measurements, slit lamp biomicroscopy, motility assessments, and vision acuity testing).
Size of Retinal Defects | From enrollment to post initial procedure at 5 years
  Annually assess the size (measured in clock hours) of retinal defects including giant retinal tears (GRT) in participants experiencing retinal defects after undergoing the OSC/SS procedure, using IDO examinations compared to the natural course of SS.
Number of Occurrences of Retinal Defects | From enrollment to post initial procedure at 5 years
  Annually assess by tracking the number of occurrences of participants experiencing retinal defects including giant retinal tears after undergoing the OSC/SS procedure, using the number of unique retinal defect forms received for each participant.
Number of Participants Experiencing Retinal Defects | From enrollment to post initial procedure at 5 years
  Annually assess by tracking the number of participants experiencing retinal defects after undergoing the OSC/SS procedure, using data from one of the following: photographic fundus mapping and IDO examinations.
Number of Surgeries to Repair Retinal Detachments or Retinal Defects | From enrollment to post initial procedure at 5 years
  Annually assess by tracking the number of surgeries to repair retinal detachments or retinal defects in participants after undergoing the OSC/SS procedure, using the number of surgeries documented on the retinal defect forms received for each participant.
Measurement of Visual Acuity in Participants with SS Before and After the OSC/SS Procedure as Assessed by Using Standard of Care Methods | From enrollment to post initial procedure at 5 years
  Impact of the OSC/SS procedure on visual acuity in participants with SS will be measured by standard of care methods including visual acuity charts and optical coherence tomography (OCT) imaging of the macula.
Number of Procedure Deviations by Treating Physicians as Assessed by Photographic Fundus Mapping | 3 to 6 months post OSC/SS procedure
  Evaluate the compliance of treating physicians in correctly performing the OSC/SS procedure on participants with SS by tracking the number of procedure deviations including protocol specified grid coverage, burn spacing, and burn intensity by conducting a central review of photographic fundus mapping.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Morris, MD, Study Director — Helen Keller Eye Research Foundation; Peter J Belin, MD, Principal Investigator — Retina Consultants of Minnesota
Locations (2):
- United States (2):
  - Retina Specialists of Alabama, Birmingham, Alabama
  - Retina Consultants of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months after publication of primary outcomes, ending 5 years following article publication.
Access Criteria: Researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  To achieve aims in the approved proposal.
  Proposals should be directed to lbeckwith@helenkellerfoundation.org. If proposals are approved after review by regulatory counsel, requestors will need to enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Background] Kim SJ, Bailey ST, Kovach JL, Lim JI, Vemulakonda GA, Ying GS, Flaxel CJ; American Academy of Ophthalmology Preferred Practice Pattern Retina/Vitreous Committee. Posterior Vitreous Detachment, Retinal Breaks, and Lattice Degeneration Preferred Practice Pattern(R). Ophthalmology. 2025 Apr;132(4):P163-P196. doi: 10.1016/j.ophtha.2024.12.023. Epub 2025 Feb 7. No abstract available. PMID 39918519
- [Background] Camp DA, Bakhsh SR, Torkashvand A, Jensen NR, Naravane AV, Belin PJ, Quiram PA, Ivanova T, Wubben TJ, Besirli CG, Bohnsack BL, Shapiro MJ, Blair MP, Hajrasouliha AR. Laser prophylaxis for retinal detachment in Stickler syndrome: A systematic review and meta-analysis. Acta Ophthalmol. 2025 Sep;103(6):e364-e373. doi: 10.1111/aos.17509. Epub 2025 May 15. PMID 40370211
- [Background] Gocuk SA, Shahzad A, Ayton L, Dawkins RCH, Ruddle JB. Paediatric glaucoma in Stickler syndromes: a comprehensive review of prevalence, comorbidities and outcomes. BMJ Open Ophthalmol. 2025 May 27;10(1):e002138. doi: 10.1136/bmjophth-2025-002138. PMID 40436442
- [Background] Fujimoto K, Nagata T, Matsushita I, Oku K, Imagawa M, Kuniyoshi K, Hayashi T, Kimoto K, Ohji M, Kusaka S, Kondo H. ULTRA-WIDE FIELD FUNDUS AUTOFLUORESCENCE IMAGING OF EYES WITH STICKLER SYNDROME. Retina. 2021 Mar 1;41(3):638-645. doi: 10.1097/IAE.0000000000002879. PMID 32639332
- [Background] Naravane AV, Belin PJ, Quiram PA. Retinal Detachment Prophylaxis for Patients With Stickler Syndrome: A Survey of Pediatric Retinal Specialist Treatment Preferences. Ophthalmic Surg Lasers Imaging Retina. 2023 Feb;54(2):102-107. doi: 10.3928/23258160-20230119-01. Epub 2023 Feb 1. PMID 36780636
- [Background] Ver Hoeve JN, Leavitt LA. Neonatal acoustically-elicited cardiac response: modulation by state and antecedent stimulation. Psychophysiology. 1985 Mar;22(2):231-6. doi: 10.1111/j.1469-8986.1985.tb01592.x. No abstract available. PMID 3991851
- [Background] Morris RE, Parma ES, Robin NH, Sapp MR, Oltmanns MH, West MR, Fletcher DC, Schuchard RA, Kuhn F. Stickler Syndrome (SS): Laser Prophylaxis for Retinal Detachment (Modified Ora Secunda Cerclage, OSC/SS). Clin Ophthalmol. 2021 Jan 6;15:19-29. doi: 10.2147/OPTH.S284441. eCollection 2021. PMID 33447008
- [Background] Fincham GS, Pasea L, Carroll C, McNinch AM, Poulson AV, Richards AJ, Scott JD, Snead MP. Prevention of retinal detachment in Stickler syndrome: the Cambridge prophylactic cryotherapy protocol. Ophthalmology. 2014 Aug;121(8):1588-97. doi: 10.1016/j.ophtha.2014.02.022. Epub 2014 May 1. PMID 24793526
- [Background] Morris RE, Kuhn F, Richardson C. Preventing Retinal Detachment: The Encircling Laser Retinopexy Technique. Clin Ophthalmol. 2023 May 30;17:1505-1513. doi: 10.2147/OPTH.S406337. eCollection 2023. PMID 37273500
- [Background] Naravane AV, Belin PJ, Pierce B, Quiram PA. Risk and Prevention of Retinal Detachments in Patients with Stickler Syndrome. Ophthalmic Surg Lasers Imaging Retina. 2022 Jan;53(1):7-11. doi: 10.3928/23258160-20211213-02. Epub 2022 Jan 1. PMID 34982001
- [Background] Khanna S, Rodriguez SH, Blair MA, Wroblewski K, Shapiro MJ, Blair MP. Laser Prophylaxis in Patients with Stickler Syndrome. Ophthalmol Retina. 2022 Apr;6(4):263-267. doi: 10.1016/j.oret.2021.11.001. Epub 2021 Nov 11. PMID 34774838
- [Background] Parma ES, Korkko J, Hagler WS, Ala-Kokko L. Radial perivascular retinal degeneration: a key to the clinical diagnosis of an ocular variant of Stickler syndrome with minimal or no systemic manifestations. Am J Ophthalmol. 2002 Nov;134(5):728-34. doi: 10.1016/s0002-9394(02)01646-x. PMID 12429250
- [Background] Morris RE, Kuhn F, Sipos T. Preventing Retinal Detachment: Where are We? Implications from Stickler Syndrome. Clin Ophthalmol. 2022 Dec 23;16:4315-4321. doi: 10.2147/OPTH.S388631. eCollection 2022. PMID 36583093
- [Background] Carroll C, Papaioannou D, Rees A, Kaltenthaler E. The clinical effectiveness and safety of prophylactic retinal interventions to reduce the risk of retinal detachment and subsequent vision loss in adults and children with Stickler syndrome: a systematic review. Health Technol Assess. 2011 Apr;15(16):iii-xiv, 1-62. doi: 10.3310/hta15160. PMID 21466760
- [Background] Ang A, Ung T, Puvanachandra N, Wilson L, Howard F, Ryalls M, Richards A, Meredith S, Laidlaw M, Poulson A, Scott J, Snead M. Vitreous phenotype: a key diagnostic sign in Stickler syndrome types 1 and 2 complicated by double heterozygosity. Am J Med Genet A. 2007 Mar 15;143A(6):604-7. doi: 10.1002/ajmg.a.31527. PMID 17318849
- [Background] Boysen KB, La Cour M, Kessel L. Ocular complications and prophylactic strategies in Stickler syndrome: a systematic literature review. Ophthalmic Genet. 2020 Jun;41(3):223-234. doi: 10.1080/13816810.2020.1747092. Epub 2020 Apr 21. PMID 32316871
- [Background] Snead MP, McNinch AM, Poulson AV, Bearcroft P, Silverman B, Gomersall P, Parfect V, Richards AJ. Stickler syndrome, ocular-only variants and a key diagnostic role for the ophthalmologist. Eye (Lond). 2011 Nov;25(11):1389-400. doi: 10.1038/eye.2011.201. Epub 2011 Sep 16. PMID 21921955
- [Background] Ang A, Poulson AV, Goodburn SF, Richards AJ, Scott JD, Snead MP. Retinal detachment and prophylaxis in type 1 Stickler syndrome. Ophthalmology. 2008 Jan;115(1):164-8. doi: 10.1016/j.ophtha.2007.03.059. Epub 2007 Aug 2. PMID 17675240
- [Background] Reddy DN, Yonekawa Y, Thomas BJ, Nudleman ED, Williams GA. Long-term surgical outcomes of retinal detachment in patients with Stickler syndrome. Clin Ophthalmol. 2016 Aug 16;10:1531-4. doi: 10.2147/OPTH.S111526. eCollection 2016. PMID 27574392
- [Background] Taylor K, Su M, Richards Z, Mamawalla M, Rao P, Chang E. Outcomes in Retinal Detachment Repair and Laser Prophylaxis for Syndromes with Optically Empty Vitreous. Ophthalmol Retina. 2023 Oct;7(10):848-856. doi: 10.1016/j.oret.2023.06.012. Epub 2023 Jun 23. PMID 37356493
- [Background] Friberg TR. Clinical experience with a binocular indirect ophthalmoscope laser delivery system. Retina. 1987 Spring;7(1):28-31. PMID 3602603
- [Background] Riffenburgh RH, Gillen DL. Statistics in medicine: Academic Press; 2020.
- [Background] Verhoekx JSN, van Etten PG, Wubbels RJ, van Meurs JC, van Overdam KA. PROPHYLACTIC LASER TREATMENT TO DECREASE THE INCIDENCE OF RETINAL DETACHMENT IN FELLOW EYES OF IDIOPATHIC GIANT RETINAL TEARS. Retina. 2020 Jun;40(6):1094-1097. doi: 10.1097/IAE.0000000000002494. PMID 30865062
- [Background] Morris RE, Sapp MR, Oltmanns MH, West MR. Correspondence. Retina. 2023 Sep 1;43(9):e52-e53. doi: 10.1097/IAE.0000000000003829. No abstract available. PMID 37141590
- [Background] Alexander P, Fincham GS, Brown S, Collins D, McNinch AM, Poulson AV, Richards A, Martin H, Wareham N, Snead MP. Cambridge Prophylactic Protocol, Retinal Detachment, and Stickler Syndrome. N Engl J Med. 2023 Apr 6;388(14):1337-1339. doi: 10.1056/NEJMc2211320. No abstract available. PMID 37018499
- [Background] Hagler WS, Crosswell HH Jr. Radial perivascular chorioretinal degeneration and retinal detachment. Trans Am Acad Ophthalmol Otolaryngol. 1968 Mar-Apr;72(2):203-16. No abstract available. PMID 5659901
- [Background] Khan AO, AlAbdi L, Patel N, Helaby R, Hashem M, Abdulwahab F, AlBadr FB, Alkuraya FS. Genetic testing results of children suspected to have Stickler syndrome type collagenopathy after ocular examination. Mol Genet Genomic Med. 2021 May;9(5):e1628. doi: 10.1002/mgg3.1628. Epub 2021 May 5. PMID 33951325
- [Background] Zauberman H, Berman ER. Measurement of adhesive forces between the sensory retina and the pigment epithelium. Exp Eye Res. 1969 Jul;8(3):276-83. doi: 10.1016/s0014-4835(69)80039-4. No abstract available. PMID 4240714
- See also: Equator Network. Consolidated Standards of Reporting Trials (CONSORT). Equator Network. 2010. Available at URL provided. Accessed November 29, 2024. — https://www.equator-network.org/reporting-guidelines/consort/
- See also: Morris R, Witherspoon CD, Kuhn F, Sapp M. Retinal detachment laser prophylaxis (by invitation). Retina Today. 2008; 2008:63-66. [Google Scholar] — https://retinatoday.com/articles/2008-mar/0308_15-php